CLINICAL TRIAL: NCT05243199
Title: Sacubitril/Valsartan for Dialysis Patients With CKD5 Stage Complicated With Hypertension- A Prospective, Randomized, Controlled Multicenter Study
Brief Title: Sacubitril/Valsartan for CKD5 Stage Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Nan Chen,MD, Principal Investigator,Director,Foreign academicians of the French National Academy of Medical Sciences,Director of institute of Nephrology affiliated to Shanghai Jiao Tong University Medical College, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (2020)(137)
Record Dates: First submitted 2022-01-19; First posted 2022-02-16 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: CKD5 Stage Dialysis; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Irbesartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): The initial dose of 50mg Qd was increased to 50mg Bid after 1 week and maintained to 100mg Bid after 2 weeks if the patient could tolerate it
  Interventions: Drug: Sacubitril/Valsartan
- Irbesartan (Active Comparator): the maximum tolerated dose of irbesartan was administered
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Sacubitril/Valsartan — The initial dose of 50mg Qd was increased to 50mg Bid after 1 week and maintained to 100mg Bid after 2 weeks if the patient could tolerate it (no follow-up exit criteria were found).
  Other Names: ARNI
  Arms: Sacubitril/Valsartan
Drug: Irbesartan — The Initial dose of 75 mg Qd with sand, such as patients can tolerate and follow-up exit criteria (not appear, to 75 mg Bid to maintain after 1 week, 2 weeks can still be tolerance is raised to 150 mg Bid.
  Other Names: ARB
  Arms: Irbesartan

SUMMARY:
Hemodialysis or peritoneal dialysis CKD5 patients were randomly divided into Sacubitril/Valsartan and irbesartan treatment groups. Comparing the blood pressure, survival rates, the cardiac function, renal function,and adverse reactions of two groups, to evaluate whether the efficacy and safety of Sacubitril/Valsartan in the treatment of patients with CKD dialysis combined with heart failure is superior to that of irbesartan.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 5, starting regular hemodialysis or peritoneal dialysis for more than 1 month.
* NT-proBNP ≥2000pg/ml.
* hypertension
* Voluntary informed consent.

Exclusion Criteria:

* Unable to tolerate ACEI/ARB class antihypertensive drugs;
* History of symptomatic hypotension/systolic blood pressure <100mmHg at screening;
* Potassium >6.0mmol/L;
* History of angioedema;
* Abnormal liver function such as ALT and/or AST >=3 times normal upper limit (ULN), total bilirubin >= 2 times ULN;
* Moderate to severe anemia (hemoglobin <80g/L);
* Cardiac surgery/intervention/cardiac resynchronization therapy has been performed in the past 3 months or is planned in the next 12 months;
* Newly found malignant tumor (within 3 years), or undergoing radiotherapy/chemotherapy;
* Pregnant and lactating women, or those of childbearing age who are unable to guarantee effective contraception;
* New and serious life-threatening infections;
* Active infectious diseases such as active tuberculosis, active viral hepatitis and HIV infection;
* Persons suffering from mental disorders and taking psychotropic drugs;
* Patients with life expectancy less than 12 months;
* The doctor assessed that the patient was not easy to follow up or had poor compliance and was not suitable for enrollment;
* Patients who do not want to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
The effect of ARNI on blood pressure in patients with CKD who are on dialysis | 1 year
  The evaluation indicator include office blood pressure

SECONDARY OUTCOMES:
The effect of ARNI on ambulatory blood pressure | 1 year
  The evaluation indicator include ambulatory blood pressure
The effect of ARNI on cardiac function in patients with CKD who are on dialysis | 1 year
  The evaluation indicators include heart function-related indicators such as NT pro-BNP and EF value
The safety of ARNI in patients with CKD who are on dialysis | 1 year
  The evaluation indicators incidence of death (including death from cardiovascular events or other causes), hyperkalemia and other adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Ruijin Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China